CLINICAL TRIAL: NCT05385731
Title: MUSCLE - Nordic and Free Walking in People With Multiple Sclerosis: Clinical-functional, Motor Control, and Gait Analysis Findings: a Randomized Controlled Multicentre Clinical Trials
Brief Title: MUSCLE - Nordic Walking in MUltiple SCLErosis
Acronym: MUSCLE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Leonardo A. Peyré-Tartaruga (Other)
Collaborators: Aline Nogueira Haas (Unknown); Flávia Gomes Martinez (Unknown)
Responsible Party: Sponsor-Investigator, Leonardo A. Peyré-Tartaruga, Associate Professor, Federal University of Rio Grande do Sul
Organization: Federal University of Rio Grande do Sul (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MUSCLE
Record Dates: First submitted 2022-02-17; First posted 2022-05-23 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Multiple Sclerosis, Chronic Progressive; Multiple Sclerosis; Multiple Sclerosis, Primary Progressive; Multiple Sclerosis, Secondary Progressive
Keywords: Mobility; Functionality; Movement disorders; Rehabilitation; Locomotion; Gait kinematics; Electromyographic activity; Quality of life
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive; Multiple Sclerosis; Movement Disorders | interventions — Nordic Walking

STUDY DESIGN:
Intervention Model Description: Study Type: Interventional, Randomized controlled multicenter clinical trial In this research, four groups of patients with Parkinson's disease will receive intervention during 4 months of different physical therapy programs (Nordic walking) and free walking, who will receive telephone guidance for performing home-based exercises. The training programs will have a duration of 4 months and will be periodized so that the duration of the sessions is matched between them. The intensity of the interval training will be manipulated by the subjective effort scale (Borg) and by the heart rate, with predetermined series durations. All training programs will have a frequency of two sessions per week and a duration of 60 minutes. In order to evaluate the effects of the training, evaluations will be performed before and after the training period: 1) Basal (month 0): initial pre-training evaluation; 2) month 4: Evaluation 48h after the last training session.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: double-blind (Investigator, Outcomes Assessor, Care Provider)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Nordic Walking (NWG) (Experimental): The Nordic Walk program consists of 3 moments:
  warm-up, walk, and stretch. They will do a brief free walking warm-up for 3 minutes in the Self-selected walking speed - SSWS (3 'SSWS), then walk according to the training cycle, the intensity will be between 60 to 80% of the Heart of Ratio reserve. In addition, the intensity of the classes will be measured in each phase by the Borg Scale of Perceived Exertion.
  Interventions: Other: Nordic Walking (NWG); Other: Free Walking (FWG); Other: Health Education (HEG)
- Free walking (FWG) (Active Comparator): The free walking program consists of 3 moments:
  warm-up, walk, and stretch. They will do a brief free walking warm-up for 3 minutes in the Self-selected walking speed - SSWS (3 'SSWS), then walk according to the training cycle, the intensity will be between 60 to 80% of the Heart of Ratio reserve. In addition, the intensity of the classes will be measured in each phase by the Borg Scale of Perceived Exertion.
  Intervention administered:
  24 sessions will be held twice a week, with each session taking an average of 60 minutes.
  Interventions: Other: Nordic Walking (NWG); Other: Free Walking (FWG); Other: Health Education (HEG)
- Health Education (HEG) (No Intervention): The control group will receive orientation and carry out the "Health Education" program and will have a duration of 3 months.

INTERVENTIONS:
Other: Nordic Walking (NWG) — 24 sessions will be held twice a week, with each session taking an average of 60 minutes.
  Arms: Free walking (FWG); Nordic Walking (NWG)
Other: Free Walking (FWG) — 24 sessions will be held twice a week, with each session taking an average of 60 minutes.
  Arms: Free walking (FWG); Nordic Walking (NWG)
Other: Health Education (HEG) — The control group will receive orientation and carry out the "Health Education" program and will have a duration of 3 months.
  Arms: Free walking (FWG); Nordic Walking (NWG)

SUMMARY:
The aim of the study is to analyze the effects of Nordic Walking and free walking in the clinical-functional, postural balance, motor control, muscular echographic quality, and gait analysis (pendulum gait mechanism), in people with Multiple Sclerosis.

DETAILED DESCRIPTION:
Objective: Analyze the effects of Nordic Walking and free walking in the clinical-functional parameters, postural balance, muscular echography quality, pendulum gait mechanism, in people with Multiple sclerosis. Experimental Design: Randomized controlled multicenter clinical trial with translational study characteristics. Search Location: Exercise Research Laboratory at the School of Physical Education, Physiotherapy and Dance, Federal University of Rio Grande do Sul, Brazil, and University of Pavia, on Department of Public Health, Experimental Medicine and Forensic Sciences, Pavia, Italy. Participants: 60 patients from the Unified Health System (UHS) of both sexes, from 20 to 75 years old, diagnosed with multiple sclerosis, sedentary. Interventions: In this research, four groups of patients with multiple sclerosis will receive intervention during 4 months of different physical therapy programs (Nordic walking and free walking), who will receive telephone guidance for performing home-based exercises. The training programs will have a duration of 3 months and will be periodized so that the duration of the sessions is matched between them. The intensity of the interval training will be manipulated by the subjective effort scale (Borg) and by the heart rate, with predetermined series durations. All training programs will have a frequency of two sessions per week and a duration of 60 minutes. To evaluate the effects of the training, evaluations will be performed before and after the training period: 1) Basal (month 0): initial pre-training evaluation; 2) month 4: Evaluation 48h after the last training session. Outcomes: clinical-functional parameters, postural balance, muscular echography quality, pendulum gait mechanism, and biochemistry. Data Analysis: Data will be described by average values and standard deviation values. The comparisons between and within groups will be performed using a Generalized Estimating Equations (GEE) analysis, adopting a level of significance (α) of 0.05. Expected Results: The intervention groups of the Nordic walking are expected to be more effective in all outcomes analyzed, especially improving functional mobility when compared to the control group of unsupervised home exercises. In addition, it is expected that the results of the research will be expandable and the possibility of future developments in the scientific, technological, economic, social, and environmental fields and that they will be implemented in the Unified Health System (UHS).

ELIGIBILITY:
Inclusion Criteria:

* volunteers aged over 20 years;
* of both sexes;
* with a clinical diagnosis of multiple sclerosis.

Exclusion Criteria:

* severe heart diseases, uncontrolled hypertension, myocardial infarction within a period of less than one year, being a pacemaker;
* stroke or other associated neurological diseases; insanity;
* prostheses in the lower limbs;
* without ambulation conditions.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-08-02 (Estimated); Primary Completion 2022-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Test Timed Up and Go | Change from baseline at 12 weeks
  Test Timed Up and Go: This test evaluates the mobility functional in three meters of self-selected speed (TUGSS) or at forced speed (TUGFS) [Time Frame: Change from baseline at 12 weeks]
Locomotor Rehabilitation Index | Change from baseline at 12 weeks
  The Locomotor Rehabilitation Index is a method of determining how close is the SSW compared to the Optimum Speed (Vopt).
Self-selected walking speed | Change from baseline at 12 weeks
  SSWS This outcome will be measure in test of treadmill walking

SECONDARY OUTCOMES:
Optimal Walking Speed (OPT) | Change from baseline at 12 weeks
  Optimal Walking Speed (OPT) This outcome will be measure through of the registered image movement analysis using the three-dimensional motion analysis system (VICON) of the walking test on treadmill.
Quality of life (QoL) | Change from baseline at 12 weeks
  Quality of life (QoL) The quality of life will be estimated using the World Health Organization Quality of Life. (WHOQOL-short domains: physical, psychological, social relationships, environment, and general quality of life) and (WHOQOL-Long domains: sensory abilities, autonomy, Past. Present and Future Activities, social participation, death and dying, intimacy, and general quality of life).
Cognitive function | Change from baseline at 12 weeks
  Cognitive function This outcome will be measure for Montreal Cognitive Assessment (MoCA).
Depressive symptoms | Change from baseline at 12 weeks
  This outcome will be measure for the Geriatric Depression Scale - 15 item. The scale consists of 15 dichotomous questions in which participants are asked to answer yes or no in reference to how they felt over the past week (for instance, "Do the patient feel that their life is empty?," Do the patient feel that their situation is hopeless?). Scores range from 0 to 15 with higher scores indicating more depressive symptoms.
Expanded Disability Status Scale | Change from baseline at 12 weeks
  The Expanded Disability Status Scale is the most appropriate to assess evolution and point to a new relapse. The Expanded Disability Status Scale has been the most commonly used. It has twenty items with scores ranging from 0 to 10, with the score increasing by half a point according to the patient's degree of disability, giving more focus on the patient's ability to walk (especially in scores above 4.0).

OTHER OUTCOMES:
Balance Dynamics | Change from baseline at 12 weeks
  Balance Dynamics: This outcome will be evaluated using Berg Balance Scale (BBS). This scale assessment of the individual's balance in 14 situations, representative of activities of the day to day, such as: stand up, get up, walk, to lean forward, to move, to turn, among others. The maximum score of a being reached of 56 points and each item has an ordinal scale of five alternatives ranging from 0 to 4 points, according to the degree of difficulty.
Balance Static | Change from baseline at 12 weeks
  Balance Static: This outcome will be evaluated using area of center of pressure (cm squared).
Stride length | Change from baseline at 12 weeks
  Stride Length (in meters). This outcome will be measure through of the registered image movement analysis using the three-dimensional motion analysis system (VICON) of the walking test on treadmill at different speed of walking (SSWS, below and above of the SSWS), 3 minutes at each speed (in kilometers/hours).
Dynamics Stability | Change from baseline at 12 weeks
  This outcome is calculated as the inter-strides variation in terms of coefficient of variation of stride frequency.
Electromyographic activity | Change from baseline at 12 weeks
  This outcome is measure is the mean amplitude (in millivolts) of the muscles: vastus lateralis (VL), biceps femoris (BF), anterior tibial (AT) and medial gastrocnemius (MG) This outcome will be measured through Measuring the electromyographic activation during treadmill walking tests using an electromyograph. In of the walking test on treadmill at different speed of walking (SSWS, below and above of the SSWS), 3 minutes at each speed.
Motor behavior by electromyographic activity | Change from baseline at 12 weeks
  During the gait initiation, the investigators will evaluate the anticipatory postural adjustments. The electromyograph will be used to obtain electromyographic activity data of the spinal erector muscles, internal oblique, gluteus medius, rectus femoris, femoral biceps, medial gastrocnemius and tibialis anterior (in mV).
  All these parameters will be measured before and after Nordic and free walking interventions.
Muscular activation | Change from baseline at 12 weeks
  Muscular activation:Muscular activation during phases of the gait cycle of people with Parkinson's disease through the electromyographic evaluation of the muscles of the spinal erector, internal oblique, gluteus medius, rectus femoris, femoral biceps, anterior tibialis and medial gastrocnemius during treadmill running. All participants will walk on a treadmill at selected walking speed. To identify electromyographic activity during the different gait cycles, the electromyograph will be synchronized with VICON (Vicon Motion Capture System - Oxford - USA, 1984).
  All these parameters will be measured before and after Nordic and free walking interventions.
Internal Work | Change from baseline at 12 weeks
  The internal work is the mechanical energy fluctuations of the movement of limbs relative to the center of body mass (Wint, in Joules). This outcome will be measured through the registered image movement analysis using the three-dimensional motion analysis system VICON of the walking test on the treadmill.
  All these parameters will be measured before and after Nordic and free walking interventions.
External Work | Change from baseline at 12 weeks
  The external work is energy fluctuations of the center of body mass with respect to the external environment or surroundings (Wext, in Joules). This outcome will be measured through the registered image movement analysis using the three-dimensional motion analysis system VICON of the walking test on the treadmill.
  All these parameters will be measured before and after Nordic and free walking interventions.
total mechanical work | Change from baseline at 12 weeks
  The total mechanical work (Wtot =Wext + Wint) produced by a body during activity. These outcomes are measured by composite for:(external, internal mechanical work, in Joules). This outcome will be measured through the registered image movement analysis using the three-dimensional motion analysis system VICON of the walking test on the treadmill.
  All these parameters will be measured before and after Nordic and free walking interventions.
Pendulum-like Recovery | Change from baseline at 12 weeks
  The mechanical energy exchange of the center of mass is quantified by the calculation of the percentage of reconversion of mechanical energy, called Recovery (R), which counts the form that the mechanical energy is saved through the pendulum mechanism of the locomotion. This outcome will be measured through the registered image movement analysis using the three-dimensional motion analysis system VICON of the walking test on the treadmill.
  This parameter will be measured before and after Nordic and free walking interventions.
Scapular and pelvis coordination | Change from baseline at 12 weeks
  The scapular girdle movement in angles will be measure, pelvic girdle in angles will be measure.
  The scapular girdle movement in angles will be aggregated to pelvic girdle in angles to arrive at continuous phases relation in angle.
  This parameter will be measured before and after Nordic and free walking interventions.
Range of motion | Change from baseline at 12 weeks
  Range of motion (in degrees) of the following segments and joints: Tilt pelvic, sagittal flexion of trunk, hip flexion, knee flexion, ankle flexion, shoulder flexion, shoulder abduction, elbow flexion. All these parameters will be measured before and after Nordic and free walking interventions.
Psychological parameters - Profile of Mood State | Change from baseline at 12 weeks
  This variable will be measure by the Brunel Mood Scale (BRUMS) that was developed to provide a quick assessment of mood states adult populations. The BRUMS has been demonstrated to have Cronbach alpha values above 0.70 and is a reliable tool used to measure the mood of Brazilian athletes. The instrument consisted of 24 items and six subscales assessing mood: tension, depression, anger, vigor, fatigue and confusion.
  Each item was rated on a Likert scale ranging from nothing (0) to extremely (4), where the respondent indicated how they were feeling at that moment. The results were calculated using the mean of the items in each subscale.
Quality of sleep - The Pittsburgh Sleep Quality Index (PSQI) | Change from baseline at 12 weeks
  The PSQI consists of 24 questions or items to be rated (0-3 for 20 items while 4 items are open-ended), 19 of which are self-reported and 5 of which require secondary feedback from a room or bed partner. Only the self-reported items (15 rated as 0-3 while 4 open-ended) are used for quantitative evaluation of sleep quality as perceived by the patient. The open-ended items are also finally scored as structured categorical values (rated at 0-3) as per the range of values reported for them by the patient. These 19 self-reported items are used to generate categorical scores representing the PSQI's 7 components. The individual component scores each assess a specific feature of sleep. Finally, the scores for each component are summed to get a total score, also termed the global score (range: 0 to 21). This score provides a summary of the respondent's sleep experience and quality for the past month.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Federal do Rio Grande do Sul, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Balbinot G, Schuch CP, Bianchi Oliveira H, Peyre-Tartaruga LA. Mechanical and energetic determinants of impaired gait following stroke: segmental work and pendular energy transduction during treadmill walking. Biol Open. 2020 Jul 21;9(7):bio051581. doi: 10.1242/bio.051581. PMID 32694152
- [Background] Baker NA, Tickle-Degnen L. The effectiveness of physical, psychological, and functional interventions in treating clients with multiple sclerosis: a meta-analysis. Am J Occup Ther. 2001 May-Jun;55(3):324-31. doi: 10.5014/ajot.55.3.324. PMID 11723974
- [Background] Cavagna GA, Thys H, Zamboni A. The sources of external work in level walking and running. J Physiol. 1976 Nov;262(3):639-57. doi: 10.1113/jphysiol.1976.sp011613. PMID 1011078
- [Background] Chung KC, Song JW; WRIST Study Group. A guide to organizing a multicenter clinical trial. Plast Reconstr Surg. 2010 Aug;126(2):515-523. doi: 10.1097/PRS.0b013e3181df64fa. PMID 20375760
- [Background] Confavreux C, Vukusic S, Adeleine P. Early clinical predictors and progression of irreversible disability in multiple sclerosis: an amnesic process. Brain. 2003 Apr;126(Pt 4):770-82. doi: 10.1093/brain/awg081. PMID 12615637
- [Background] Correale L, Buzzachera CF, Liberali G, Codrons E, Mallucci G, Vandoni M, Montomoli C, Bergamaschi R. Effects of Combined Endurance and Resistance Training in Women With Multiple Sclerosis: A Randomized Controlled Study. Front Neurol. 2021 Aug 5;12:698460. doi: 10.3389/fneur.2021.698460. eCollection 2021. PMID 34421801
- [Background] Dos Santos Delabary M, Monteiro EP, Donida RG, Wolffenbuttel M, Peyre-Tartaruga LA, Haas AN. Can Samba and Forro Brazilian rhythmic dance be more effective than walking in improving functional mobility and spatiotemporal gait parameters in patients with Parkinson's disease? BMC Neurol. 2020 Aug 18;20(1):305. doi: 10.1186/s12883-020-01878-y. PMID 32811464
- [Background] Detrembleur C, van den Hecke A, Dierick F. Motion of the body centre of gravity as a summary indicator of the mechanics of human pathological gait. Gait Posture. 2000 Dec;12(3):243-50. doi: 10.1016/s0966-6362(00)00081-3. PMID 11154935
- [Background] Gomenuka NA, Oliveira HB, da Silva ES, Passos-Monteiro E, da Rosa RG, Carvalho AR, Costa RR, Rodriguez Paz MC, Pellegrini B, Peyre-Tartaruga LA. Nordic walking training in elderly, a randomized clinical trial. Part II: Biomechanical and metabolic adaptations. Sports Med Open. 2020 Jan 13;6(1):3. doi: 10.1186/s40798-019-0228-6. PMID 31932999
- [Background] Kalb R, Brown TR, Coote S, Costello K, Dalgas U, Garmon E, Giesser B, Halper J, Karpatkin H, Keller J, Ng AV, Pilutti LA, Rohrig A, Van Asch P, Zackowski K, Motl RW. Exercise and lifestyle physical activity recommendations for people with multiple sclerosis throughout the disease course. Mult Scler. 2020 Oct;26(12):1459-1469. doi: 10.1177/1352458520915629. Epub 2020 Apr 23. PMID 32323606
- [Background] MONTEIRO, Elren Passos et al. Aspectos biomecânicos da locomoção de pessoas com doença de Parkinson: revisão narrativa. Revista Brasileira de Ciências do Esporte, v. 39, p. 450-457, 2017.
- [Background] Motl RW, Sandroff BM. Benefits of Exercise Training in Multiple Sclerosis. Curr Neurol Neurosci Rep. 2015 Sep;15(9):62. doi: 10.1007/s11910-015-0585-6. PMID 26223831
- [Background] O'CONNELL, R. et al. A controlled study to assess the effects of aerobic training on patients with multiple sclerosis. 14th International World Confederation for Physical Therapy, 2003.
- [Background] Passos-Monteiro E, B Schuch F, T Franzoni L, R Carvalho A, A Gomenuka N, Becker M, Rieder CRM, Andrade A, G Martinez F, S Pagnussat A, A Peyre-Tartaruga L. Nordic Walking and Free Walking Improve the Quality of Life, Cognitive Function, and Depressive Symptoms in Individuals with Parkinson's Disease: A Randomized Clinical Trial. J Funct Morphol Kinesiol. 2020 Nov 10;5(4):82. doi: 10.3390/jfmk5040082. PMID 33467297
- [Background] Patti F, Ciancio MR, Cacopardo M, Reggio E, Fiorilla T, Palermo F, Reggio A, Thompson AJ. Effects of a short outpatient rehabilitation treatment on disability of multiple sclerosis patients--a randomised controlled trial. J Neurol. 2003 Jul;250(7):861-6. doi: 10.1007/s00415-003-1097-x. PMID 12883930
- [Background] Peyre-Tartaruga LA, Martinez FG, Zanardi APJ, Casal MZ, Donida RG, Delabary MS, Passos-Monteiro E, Coertjens M, Haas AN. Samba, deep water, and poles: a framework for exercise prescription in Parkinson's disease. Sport Sci Health. 2022;18(4):1119-1127. doi: 10.1007/s11332-022-00894-4. Epub 2022 Feb 17. PMID 35194464
- [Background] Polman CH, Reingold SC, Banwell B, Clanet M, Cohen JA, Filippi M, Fujihara K, Havrdova E, Hutchinson M, Kappos L, Lublin FD, Montalban X, O'Connor P, Sandberg-Wollheim M, Thompson AJ, Waubant E, Weinshenker B, Wolinsky JS. Diagnostic criteria for multiple sclerosis: 2010 revisions to the McDonald criteria. Ann Neurol. 2011 Feb;69(2):292-302. doi: 10.1002/ana.22366. PMID 21387374
- [Background] Psarakis M, Greene D, Moresi M, Baker M, Stubbs P, Brodie M, Lord S, Hoang P. Impaired heel to toe progression during gait is related to reduced ankle range of motion in people with Multiple Sclerosis. Clin Biomech (Bristol). 2017 Nov;49:96-100. doi: 10.1016/j.clinbiomech.2017.08.012. Epub 2017 Sep 1. PMID 28898816
- [Background] Rietberg MB, Brooks D, Uitdehaag BM, Kwakkel G. Exercise therapy for multiple sclerosis. Cochrane Database Syst Rev. 2005 Jan 25;2005(1):CD003980. doi: 10.1002/14651858.CD003980.pub2. PMID 15674920
- [Background] Schepens B, Bastien GJ, Heglund NC, Willems PA. Mechanical work and muscular efficiency in walking children. J Exp Biol. 2004 Feb;207(Pt 4):587-96. doi: 10.1242/jeb.00793. PMID 14718502
- [Background] SOARES, Gustavo da Silva; PEYRÉ-TARTARUGA, Leonardo Alexandre. Doença de Parkinson e exercício físico: uma revisão da literatura. Ciência em Movimento, v. 12, n. 24, p. 69-85, 2010.
- [Background] Reuter I, Mehnert S, Leone P, Kaps M, Oechsner M, Engelhardt M. Effects of a flexibility and relaxation programme, walking, and nordic walking on Parkinson's disease. J Aging Res. 2011;2011:232473. doi: 10.4061/2011/232473. Epub 2011 Mar 30. PMID 21603199
- [Background] Tschentscher M, Niederseer D, Niebauer J. Health benefits of Nordic walking: a systematic review. Am J Prev Med. 2013 Jan;44(1):76-84. doi: 10.1016/j.amepre.2012.09.043. PMID 23253654
- [Background] YASINSKAYA, Yana Konstantinovna. DEVELOPMENT OF STATIC AND DYNAMIC BALANCE IN INDIVIDUALS WITH MULTIPLE SCLEROSIS BASED ON THE USE OF THE NORDIC WALKING METHOD. имени ПФ Лесгафта, n. 12, p. 320, 2014.
- [Background] WILLEMS, P.-A.; SCHEPENS, Bénédicte; DETREMBLEUR, Christine. Marcha normal. EMC-Kinesiterapia-Medicina Física, v. 33, n. 2, p. 1-29, 2012.
- [Background] Zanardi APJ, da Silva ES, Costa RR, Passos-Monteiro E, Dos Santos IO, Kruel LFM, Peyre-Tartaruga LA. Gait parameters of Parkinson's disease compared with healthy controls: a systematic review and meta-analysis. Sci Rep. 2021 Jan 12;11(1):752. doi: 10.1038/s41598-020-80768-2. PMID 33436993
- [Result] Boeschoten RE, Braamse AMJ, Beekman ATF, Cuijpers P, van Oppen P, Dekker J, Uitdehaag BMJ. Prevalence of depression and anxiety in Multiple Sclerosis: A systematic review and meta-analysis. J Neurol Sci. 2017 Jan 15;372:331-341. doi: 10.1016/j.jns.2016.11.067. Epub 2016 Nov 30. PMID 28017241
- [Result] Casal MZ, Peyre-Tartaruga LA, Zanardi APJ, Ivaniski-Mello A, Alves LL, Haas AN, Martinez FG. Postural Adjustments and Biomechanics During Gait Initiation and Obstacle Negotiation: A Comparison Between Akinetic-Rigid and Hyperkinetic Parkinson's Disease. Front Physiol. 2021 Nov 4;12:723628. doi: 10.3389/fphys.2021.723628. eCollection 2021. PMID 34803726
- [Result] Cavagna GA, Willems PA, Legramandi MA, Heglund NC. Pendular energy transduction within the step in human walking. J Exp Biol. 2002 Nov;205(Pt 21):3413-22. doi: 10.1242/jeb.205.21.3413. PMID 12324550
- [Result] Frazzitta G, Balbi P, Maestri R, Bertotti G, Boveri N, Pezzoli G. The beneficial role of intensive exercise on Parkinson disease progression. Am J Phys Med Rehabil. 2013 Jun;92(6):523-32. doi: 10.1097/PHM.0b013e31828cd254. PMID 23552330
- [Result] Gomenuka NA, Bona RL, da Rosa RG, Peyre-Tartaruga LA. The pendular mechanism does not determine the optimal speed of loaded walking on gradients. Hum Mov Sci. 2016 Jun;47:175-185. doi: 10.1016/j.humov.2016.03.008. Epub 2016 Mar 24. PMID 27017543
- [Result] Gulde P, Hermsdorfer J, Rieckmann P. Speed but Not Smoothness of Gait Reacts to Rehabilitation in Multiple Sclerosis. Mult Scler Int. 2021 Jun 3;2021:5589562. doi: 10.1155/2021/5589562. eCollection 2021. PMID 34123427
- [Result] Halabchi F, Alizadeh Z, Sahraian MA, Abolhasani M. Exercise prescription for patients with multiple sclerosis; potential benefits and practical recommendations. BMC Neurol. 2017 Sep 16;17(1):185. doi: 10.1186/s12883-017-0960-9. PMID 28915856
- [Result] Hobart JC, Riazi A, Lamping DL, Fitzpatrick R, Thompson AJ. Measuring the impact of MS on walking ability: the 12-Item MS Walking Scale (MSWS-12). Neurology. 2003 Jan 14;60(1):31-6. doi: 10.1212/wnl.60.1.31. PMID 12525714
- [Result] Kelleher KJ, Spence W, Solomonidis S, Apatsidis D. The characterisation of gait patterns of people with multiple sclerosis. Disabil Rehabil. 2010;32(15):1242-50. doi: 10.3109/09638280903464497. PMID 20156050
- [Result] Kim Y, Lai B, Mehta T, Thirumalai M, Padalabalanarayanan S, Rimmer JH, Motl RW. Exercise Training Guidelines for Multiple Sclerosis, Stroke, and Parkinson Disease: Rapid Review and Synthesis. Am J Phys Med Rehabil. 2019 Jul;98(7):613-621. doi: 10.1097/PHM.0000000000001174. PMID 30844920
- [Result] Kuo AD, Donelan JM. Dynamic principles of gait and their clinical implications. Phys Ther. 2010 Feb;90(2):157-74. doi: 10.2522/ptj.20090125. Epub 2009 Dec 18. PMID 20023002
- [Result] Kurtzke JF. Rating neurologic impairment in multiple sclerosis: an expanded disability status scale (EDSS). Neurology. 1983 Nov;33(11):1444-52. doi: 10.1212/wnl.33.11.1444. PMID 6685237
- [Result] Leal-Nascimento AH, da Silva ES, Zanardi APJ, Ivaniski-Mello A, Passos-Monteiro E, Martinez FG, Rodrigo de Carvalho A, Baptista RR, Peyre-Tartaruga LA. Biomechanical responses of Nordic walking in people with Parkinson's disease. Scand J Med Sci Sports. 2022 Feb;32(2):290-297. doi: 10.1111/sms.14095. Epub 2021 Dec 7. PMID 34780079
- [Result] Martinez-Lemos I, Martinez-Aldao D, Seijo-Martinez M, Ayan C. Nordic walking for people with relapsing-remittent multiple sclerosis: A case series study. Mult Scler Relat Disord. 2020 Nov;46:102479. doi: 10.1016/j.msard.2020.102479. Epub 2020 Sep 3. PMID 32911307
- [Result] Nardello F, Ardigo LP, Minetti AE. Measured and predicted mechanical internal work in human locomotion. Hum Mov Sci. 2011 Feb;30(1):90-104. doi: 10.1016/j.humov.2010.05.012. Epub 2010 Nov 5. PMID 21056491
- [Result] Nogueira LA, Teixeira L, Sabino P, Filho HA, Alvarenga RM, Thuler LC. Gait characteristics of multiple sclerosis patients in the absence of clinical disability. Disabil Rehabil. 2013 Aug;35(17):1472-8. doi: 10.3109/09638288.2012.738760. PMID 23869824
- [Result] Peyre-Tartaruga LA, Dewolf AH, di Prampero PE, Fabrica G, Malatesta D, Minetti AE, Monte A, Pavei G, Silva-Pereyra V, Willems PA, Zamparo P. Mechanical work as a (key) determinant of energy cost in human locomotion: recent findings and future directions. Exp Physiol. 2021 Sep;106(9):1897-1908. doi: 10.1113/EP089313. Epub 2021 Jul 14. PMID 34197674
- [Result] Proschinger S, Kuhwand P, Rademacher A, Walzik D, Warnke C, Zimmer P, Joisten N. Fitness, physical activity, and exercise in multiple sclerosis: a systematic review on current evidence for interactions with disease activity and progression. J Neurol. 2022 Jun;269(6):2922-2940. doi: 10.1007/s00415-021-10935-6. Epub 2022 Jan 27. PMID 35084560
- [Result] Saibene F, Minetti AE. Biomechanical and physiological aspects of legged locomotion in humans. Eur J Appl Physiol. 2003 Jan;88(4-5):297-316. doi: 10.1007/s00421-002-0654-9. Epub 2002 Nov 13. PMID 12527959
- [Result] Zigmond MJ, Smeyne RJ. Exercise: is it a neuroprotective and if so, how does it work? Parkinsonism Relat Disord. 2014 Jan;20 Suppl 1:S123-7. doi: 10.1016/S1353-8020(13)70030-0. PMID 24262162